CLINICAL TRIAL: NCT03801122
Title: Study of Thromboelastography During Tranexamic Acid Treatment in Preventing Bleeding in Patients With Haematological Malignancies Presenting Severe Thrombocytopenia (TTRAP-bleeding)
Brief Title: Evolution of Thromboelastography During Tranexamic Acid Treatment
Acronym: TTRAP-Bleeding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-1201; 2018-004756-38 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2019-01-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hematological Malignancies Treated With Intensive Chemotherapy
Keywords: Tranexamic acid; bleeding; hematological malignancies; thrombocytopenia
MeSH Terms: conditions — Hemorrhage; Hematologic Neoplasms; Thrombocytopenia | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Arm 1 : Tranexamic acid 3g/day Arm 2 : Tranexamic acid 1.5g/day Arm 3 : No tranexamic acid
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tranexamic acid 3g/day (Experimental): Administration of tranexamic acid 3g/day, with 3 injections/8 hours.
  Interventions: Drug: Tranexamic acid
- Tranexamic acid 1.5g/day (Experimental): Administration of tranexamic acid 1.5g/day, with 3 injections/8 hours.
  Interventions: Drug: Tranexamic acid
- No treatment (No Intervention): No treatment (no administration of tranexamic acid)

INTERVENTIONS:
Drug: Tranexamic acid — Administration of tranexamic acid, with 3 injections/8 hours.
  Arms: Tranexamic acid 1.5g/day; Tranexamic acid 3g/day

SUMMARY:
Patients with hematological malignancies are at increased risk of bleeding, especially during intensive chemotherapy. The aim of this study is to compare by thromboelastography changes during the intensive chemotherapy in patients with hematological malignancies.

DETAILED DESCRIPTION:
Patients with hematological malignancies often develop low platelet counts either as a consequence of the disease or the treatment by chemotherapy or stem cell transplantation. Platelet transfusions are commonly given to raise any low platelet count and reduce the risk of clinical bleeding (prophylaxis) or stop active bleeding (therapy). The last studies have showed that many patients continue to experience bleeding, despite the use of platelet transfusions. Tranexamic acid is an antifibrinolytic agent. It reduces the breakdown of clots formed. This treatment is widely used in medicine (e.g. emergency, surgery, post-partum) and decreases blood loss and the use of red cell transfusions. The purpose of this study is to test different doses of tranexamic acid (full dose: 3g/day and half dose (1.5g/day) and to study its effect by thromboelastography, with the aim to determine the optimal posology for further clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security regimen or beneficiary of the same
* Signed written informed consent form
* Confirmed diagnosis of a hematological malignancy and undergoing intensive chemotherapy
* Expected to experience hypoproliferative thrombocytopenia resulting in a platelet count of ≤10 G/L for ≥ 5 days

Exclusion Criteria:

* Pregnant women
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent
* Refractoriness to platelet transfusion or requirement for a specific type of platelet transfusion (ABO-compatible, plasma-free)
* Ongoing anticoagulant therapy or antiplatelet therapy at the time of enrolment
* Treatment with any pro-coagulant agent within 48 hours of enrolment, or enrolment in other trials involving platelet transfusions, platelet growth factors, or presentation of a known hypercoagulable state
* Diagnosis of arterial or venous thromboembolic disease within the previous year
* Patient experiencing a bleeding event WHO grade ≥ 2 within 7 days before inclusion
* contra-indications to tranexamic acid (allergy, history of seizures, creatinine clearance < 30 mL/min)
* Refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Level of amplitude observed in thromboelastography | 30 days
  Amplitude levels observed in thromboelastography will be reported

SECONDARY OUTCOMES:
Time at the beginning of the clot | 30 minutes
  Time at the beginning of the clot will be reported in minutes
Clot formation time | 30 minutes
  Clot formation time will ne reported in minutes
Alpha angle | 30 days
  Alpha angle will be measured in degrees
Percentage of lysis after 30min | 30 minutes
  Percentage of lysis after 30min will be measured
Proportion of patients experiencing bleeding of WHO (World Health Organisation ) grade 2 or above | 30 days
  Proportion of patients experiencing bleeding of WHO (World Health Organisation ) grade 2 or above will be reported
Number of adverse events | 3 months
  Number of adverse events will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Chalayer, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No